CLINICAL TRIAL: NCT02324920
Title: Benefit of Dual-chamber Pacing With Closed Loop Stimulation (CLS) in Tilt-induced Cardioinhibitory Reflex Syncope. A Randomized Double-blind Parallel Trial.
Brief Title: Benefit of Dual-chamber Pacing With Closed Loop Stimulation (CLS) in Tilt-induced Cardioinhibitory Reflex Syncope
Acronym: BIOSync CLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BA103
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2020-07

CONDITIONS: Syncope
Keywords: Syncope; Closed Loop Stimulation; CLS
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DDD+CLS (Experimental): The pacemaker will be programmed in a dual-chamber DDD pacing mode with the Closed Loop Stimulation (CLS) function ON.
  Interventions: Device: DDD-CLS
- ODO (Placebo Comparator): The pacemaker will be programmed in ODO mode.
  Interventions: Device: ODO

INTERVENTIONS:
Device: DDD-CLS
  Arms: DDD+CLS
Device: ODO
  Arms: ODO

SUMMARY:
The purpose of this study is to assess whether the Closed Loop Stimulation (CLS) in addition to the DDD pacing is effective in reducing syncopal recurrences. The study hypothesis is that DDD pacing with CLS stimulation is able to prevent syncopal recurrences completely or partially by transforming syncope in pre-syncope.

ELIGIBILITY:
Inclusion Criteria:

Patients affected by clinical diagnosis of reflex syncope who meet all the following criteria:

* age >=40 years
* significant limitation of social and working life due to unpredictable or frequent syncope recurrences, ≥2 within the last year.
* type 2B cardio-inhibitory response to TT (according to the VASIS classification).
* Alternative therapies have failed or were not feasible.
* exclusion of other possible competitive causes of syncope.

Exclusion Criteria:

- Any other indication to IPG, implantable defibrillator (ICD), cardiac resynchronization therapy (CRT), according to current guidelines

Any cardiac dysfunctions possibly leading to loss of consciousness:

* overt heart failure;
* ejection fraction (LVEF) <40% (Echo-assessed within 3-month prior to study participation);
* myocardial infarction;
* diagnosis of hypertrophic or dilated cardiomyopathy;
* clinically significant valvular disease;
* sinus bradycardia <50 bpm or sinoatrial block;
* Mobitz I second-degree atrioventricular block;
* Mobitz II second or third-degree atrioventricular block;
* bundle-branch block;
* rapid paroxysmal supraventricular tachycardia or ventricular tachycardia;
* preexcited QRS complexes;
* prolonged QT interval;
* Brugada syndrome;
* arrhythmogenic right ventricular cardiomyopathy
* Symptomatic orthostatic hypotension diagnosed by standing BP measurement;
* Nonsyncopal loss of consciousness (eg, epilepsy, psychiatric, metabolic, drop-attack, cerebral transient ischemic attack, intoxication, cataplexy).
* Symptomatic cardioinhibitory carotid sinus hypersensitivity.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- CHUS Sherbrooke, Sherbrooke, Canada
- France (3):
  - Pais d'Aix, Aix-en-Provence
  - Hopital de la Timone, Marseille
  - Clinique Pasteur, Toulouse
- Italy (12):
  - Azienda Ospedaliera Pia Fondazione di Culto e Religione Cardinale G. Panico, Tricase, BA
  - Policlinico Consorziale, Bari
  - Ospedale Centrale di Bolzano, Bolzano
  - A.O. Pugliese-Ciaccio, Catanzaro
  - Ospedale San Martino, Genova
  - Azienda Ospedaliera Niguarda Ca' Granda, Milan
  - A.O. Dei Colli - Monaldi - University of Campania "Luigi Vanvitelli", Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - A.O.U. San Luigi Gonzaga, Orbassano
  - AO di Parma, Parma
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Policlinico Casilino, Roma
- Netherlands (3):
  - AMC Academic Medical Center, Amsterdam
  - Rijnstate Ziekenjuis, Arnhem
  - Zuyderland Medisch Centrum, Heerlen
- Santa Marta, Lisbon, Portugal
- Spain (4):
  - Hospital De Bellvitge, Barcelona
  - Hospital Universitario Vall d'Hebròn, Barcelona
  - Hospital Universitario Nuestra Senora de la Candelaria, Santa Cruz
  - Hospital Virgen del Rocio, Seville

REFERENCES:
- [Derived] Brignole M, Russo V, Arabia F, Oliveira M, Pedrote A, Aerts A, Rapacciuolo A, Boveda S, Deharo JC, Maglia G, Nigro G, Giacopelli D, Gargaro A, Tomaino M; BioSync CLS trial Investigators. Cardiac pacing in severe recurrent reflex syncope and tilt-induced asystole. Eur Heart J. 2021 Feb 1;42(5):508-516. doi: 10.1093/eurheartj/ehaa936. PMID 33279955
- [Derived] Brignole M, Tomaino M, Aerts A, Ammirati F, Ayala-Paredes FA, Deharo JC, Del Rosso A, Hamdan MH, Lunati M, Moya A, Gargaro A; BIOSync Study Steering Committee. Benefit of dual-chamber pacing with Closed Loop Stimulation in tilt-induced cardio-inhibitory reflex syncope (BIOSync trial): study protocol for a randomized controlled trial. Trials. 2017 May 4;18(1):208. doi: 10.1186/s13063-017-1941-4. PMID 28472974

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Pacing (DDD+CLS): The pacemaker will be programmed in a dual-chamber DDD pacing mode with the Closed Loop Stimulation (CLS) function ON.
  DDD-CLS
- Inactive Pacing (ODO): The pacemaker will be programmed in ODO mode.
  ODO
Period: Overall Study
Arm/Group | Active Pacing (DDD+CLS) | Inactive Pacing (ODO)
Started | 64 | 64
Completed | 63 | 64
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Pacing (DDD+CLS) | Inactive Pacing (ODO) | Total
Number analyzed (Participants) | 63 | 64 | 127
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [54 to 70] | 63 [56 to 73] | 63 [56 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 27 | 45
  Male | 45 | 37 | 82
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 63 | 64 | 127

OUTCOME MEASURES:

1. Primary Outcome: Patients With Recurrence of Syncopal Episode
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pacing (DDD+CLS) | Inactive Pacing (ODO)
Number analyzed (Participants) | 63 | 64
Participants | 10 | 34
Statistical Analysis 1: Comparison: Active Pacing (DDD+CLS) vs Inactive Pacing (ODO); Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.22, 95% CI 2-sided [0.11 to 0.46]; Additional models were implemented to control for country and investigational sites effect on primary endpoint

2. Secondary Outcome: Patients With Recurrence of Pre-syncope or Syncope
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active Pacing (DDD+CLS) | Inactive Pacing (ODO)
Number analyzed (Participants) | 63 | 64
Participants | 24 | 40
Statistical Analysis 1: Comparison: Active Pacing (DDD+CLS) vs Inactive Pacing (ODO); Test type: Superiority; p = 0.002, Regression, Cox; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.27 to 0.75]

ADVERSE EVENTS:
Time Frame: median follow-up period of 14.1 months
Arm/Group | Active Pacing (DDD+CLS) | Inactive Pacing (ODO)
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 4/64 | 4/64
Other Adverse Events (participants affected / at risk) | 20/64 | 39/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Pacing (DDD+CLS) (N=64) | Inactive Pacing (ODO) (N=64)
Subtalar arthrodesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
inguinal hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
NSTEMI (Cardiac disorders) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 1 (1)
pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
lead dislodgement (Cardiac disorders) | 1 (1) | 0 (0)
lead was not properly connected to the pacemaker (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Pacing (DDD+CLS) (N=64) | Inactive Pacing (ODO) (N=64)
syncope (Nervous system disorders) | 10 (10) | 33 (33)
presyncope (Cardiac disorders) | 5 (5) | 2 (2)
Keloid formation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
mild pocket bleeding (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
unspecified pain around the chest/ pocket. (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
palpitations (Cardiac disorders) | 1 (1) | 0 (0)
inappropriate pacing due to undersensing (Cardiac disorders) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 1 (1) | 1 (1)
incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
fatigue (mild obstructive sleep apnea syndrome) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT02324920/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT02324920/SAP_001.pdf